CLINICAL TRIAL: NCT01649947
Title: Modulation of Autophagy With Hydroxychloroquine in Patients With Advanced/Recurrent Non-small Cell Lung Cancer - a Phase II Study. A Study of The Cancer Institute of New Jersey Oncology Group (CINJOG)
Brief Title: Modulation of Autophagy in Patients With Advanced/Recurrent Non-small Cell Lung Cancer - Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0220110249; 0220110249 (Other: UMDNJ IRB Number); P30CA072720 (NIH); NCI-2011-03731 (Other: CTRP (Clinical Trials Reporting System)); 031105 (Other: Rutgers Cancer Institute of New Jersey)
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2022-11-21 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer; Advanced Non-small Cell Lung Cancer; Recurrent Non-small Cell Lung Cancer
Keywords: Lung cancer; Non-small cell lung cancer; Advanced non-small cell lung cancer; Recurrent non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Paclitaxel; Carboplatin; Hydroxychloroquine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 2: Bevacizumab ineligible patients (Experimental): Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Hydroxychloroquine 200 mg PO BID
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Hydroxychloroquine
- Cohort 1: Bevacizumab eligible patients (Experimental): Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Bevacizumab 15 mg/kg IV over 90 min for Hydroxychloroquine 200 mg PO BID
  Interventions: Drug: Paclitaxel; Drug: Carboplatin; Drug: Hydroxychloroquine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel will be given at a dose of 200 mg/m2(by IV over 3 hours on Day 1). Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Other Names: Taxol
Drug: Carboplatin — Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Other Names: Paraplatin
Drug: Hydroxychloroquine — Hydroxychloroquine will be given as a flat dose of 200 mg orally BID (total daily dose of 400 mg). Cycles every 3 weeks for 4-6 Cycles.
  Other Names: Plaquenil
Drug: Bevacizumab — Cohort 1 only:
  Bevacizumab will be given by IV on Day 1 of each 21-day cycle at a dose of 15 mg/kg. Cycles every 3 weeks for 4-6 Cycles.
  Other Names: Avastin
  Arms: Cohort 1: Bevacizumab eligible patients

SUMMARY:
The purpose of this study is to examine the combination of one standard treatment for lung cancer plus an additional drug, hydroxychloroquine. The standard treatment for lung cancer being used includes 2 chemotherapy drugs, called paclitaxel and carboplatin. Some patients who have a specific type of lung cancer can also receive another drug, a drug that targets blood vessels, called bevacizumab (also known as avastin). Hydroxychloroquine is an FDA approved drug for the treatment of malaria, rheumatoid arthritis and lupus erythematosis.

ELIGIBILITY:
Inclusion Criteria:

* Signed a protocol-specific informed consent.
* 18 years of age or older.
* ECOG Performance Status 0 or 1.

Cancer criteria:

* Histologically or cytologically confirmed non-small cell lung cancer. Mixed tumors will be categorized by the predominant cell type unless small cell elements are present, in which case the patient is ineligible. Cytologic or histologic elements can be established on metastatic tumor aspirate or biopsy. Sputum cytology alone is not sufficient.
* Advanced stage NSCLC (stage IVa ((malignant pleural effusion (is now staged as stage IVa by the most recent staging system), or stage IV, or recurrent disease)).
* Measurable disease according to RECIST criteria.
* Patient with CNS metastasis are required to have stable disease documented by being off treatment (surgery, or Whole Brain radiation therapy) for at least 2 weeks, and four (4) weeks is preferred. No delay in onset of therapy is required for those patients who undergo stereotactic RT to the brain lesion(s). A contrast enhanced brain CT or brain MRI is required within 35 days of enrollment. Patients with brain metastases who qualify for protocol therapy will be included in Cohort 2 (ineligible for treatment with Bevacizumab).
* Prior radiation to sites other than the brain is allowed, if completed at least 2 weeks before treatment and provided that all radiation-related toxicities have resolved to ≤ Grade 1. Stereotactic irradiation to any site excludes the need for a waiting period.

Laboratory requirements

- Adequate organ function, as evidenced by ALL the following:

* absolute neutrophil count (ANC) ≥ 1500/mm³
* platelet count ≥ 100,000/mm³
* hemoglobin ≥ 9 gm/dL
* total bilirubin ≤ 1.5 x ULN; if patient has Gilbert's disease, then patient must have isolated hyperbilirubinemia (e.g. no other liver function test abnormality), with maximum bilirubin ≤ 2 X institutional ULN.
* AST and ALT ≤ 2.5 x ULN in the absence of liver metastases; AST and ALT ≤ 5 x ULN in the presence of liver metastases
* alkaline phosphatase ≤ 2.5 x ULN
* creatinine ≤ 1.5 X institutional ULN or calculated creatinine clearance ≥ 60 ml/min as estimated using the Cockcroft-Gault formula.

Comorbidities For Cohort 1: (Bevacizumab eligible)

* For patients who have had a major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to enrollment, or anticipate the need for such while on active treatment, may participate and receive Bevacizumab at the start of the second or third cycle as they would under standard care. Placement of vascular access device is not considered major surgery, but the incision must have healed before initiation of treatment.
* Patients must have a systolic blood pressure ≤ 150 mm Hg and diastolic blood pressure ≤ 100 mm Hg (the use of antihypertensive medications to achieve these goals is allowed).
* Adequate organ function

  * INR ≤ 1.5 and aPTT WNL.
  * Urine Protein Creatinine (UPC) ratio < 1.0 or 24 hour urine protein ratio < 1000 mg

UPC ratio of spot urine is an estimation of the 24 urine protein excretion. A UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1 gm. To obtain a UPC ratio:

* Obtain at least 4 mL of a random urine sample
* Determine protein and creatinine concentration
* Calculate the UPC using one of the following formulae [urine protein]/[urine creatinine] - if both values are reported in mg/dL [(urine protein) x 0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L

For ALL (Cohort 1 and Cohort 2):

* Women must:

  * Have a negative serum or urine pregnancy test within 7 days prior to study entry if she is a woman of child-bearing potential, OR
  * Be at least one year post-menopausal, OR
  * Be surgically sterile
* Patients of childbearing or child fathering potential must be willing to use an acceptable method of birth control prior to study entry and for the duration of the study. Acceptable methods of contraception include hormonal, barrier methods, intrauterine device, tubal ligation/vasectomy or abstinence.

Exclusion Criteria:

Cancer criteria:

* No prior cytotoxic chemotherapy or targeted therapy in the advanced or metastatic setting. Post-operative adjuvant therapy for previously resected NSCLC is allowed as long as the last dose was given greater than 1 year before study entry, and there is current evidence of disease progression.
* No active malignancy other than NSCLC. Patients with a history of basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, or ductal or lobular carcinoma in situ of the breast within the past 3 years must have been treated with curative intent. Patients with a history of prior malignancy are eligible provided they were treated with curative intent and have been free of disease for > 3 years.

Comorbidities

For Cohort 1: (Bevacizumab eligible)

* No history of gross hemoptysis (defined as bright red blood of a half-teaspoon or more) within 3 months prior to enrollment.
* None of the following conditions within 6 months prior to enrollment: myocardial infarction, stroke or symptomatic peripheral vascular disease.
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to enrollment.
* No serious non-healing wound, ulcer or bone fracture.
* Patients must not have unstable angina or NYHA classification of congestive heart failure of Grade ≥ 2.
* No history of significant vascular disease (eg aortic aneurysm).
* No current or recent (within 28 days of enrollment) full dose anticoagulants or thrombolytic agents.

For Cohort 2 (Bevacizumab ineligible):

* None of the following conditions within 6 months prior to enrollment: myocardial infarction, stroke or symptomatic peripheral vascular disease.
* Patients must not have unstable angina or NYHA classification of congestive heart failure of Grade ≥ 2.
* No history of significant vascular disease (eg aortic aneurysm).

For ALL (Cohort 1 and Cohort 2):

* Patients must not have psoriasis or porphyria.
* No known hypersensitivity to 4-aminoquinoline compound.
* Patients must not have known or suspected G-6P deficiency.
* No know bleeding diathesis or coagulopathy.
* No known GI pathology that would interfere with drug bioavailability.
* No peripheral or sensory neuropathy > Grade 1 at study entry.
* No known prior hypersensitivity to carboplatin, paclitaxel, bevacizumab or hydroxychloroquine or any of their components.
* No ongoing or active infection at study entry.
* Patients must not be receiving treatment for rheumatoid arthritis or systemic lupus erythematosus.
* Patients must not have HIV or be taking HAART therapy.
* Patients must not have a history of any condition (social or medical) that, in the opinion of the Investigator, might interfere with the patient's compliance with the protocol or pose additional or unacceptable risk to the patient.
* Women must NOT be pregnant or breastfeeding.
* Must not be taking hydroxychloroquine for treatment or prophylaxis of malaria.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2011-12-23 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Aisner, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - Robert Wood Johnson University Hospital at Hamilton, Hamilton, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey Oncology Group. The study was open to accrual on 12/23/2011 and closed to accrual on 06/30/2015.
Pre-assignment Details: We are reporting results on 32 eligible patients. Seven patients were deemed ineligible.
Groups:
- Cohort 1: Bevacizumab Eligible Patients: Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Bevacizumab 15 mg/kg IV over 90 min for Hydroxychloroquine 200 mg PO BID
  Paclitaxel: Paclitaxel will be given at a dose of 200 mg/m2(by IV over 3 hours on Day 1).
  Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Carboplatin: Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Hydroxychloroquine: Hydroxychloroquine will be given as a
- Cohort 2: Bevacizumab Ineligible Patients: Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Hydroxychloroquine 200 mg PO BID
  Paclitaxel: Paclitaxel will be given at a dose of 200 mg/m2(by IV over 3 hours on Day 1).
  Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Carboplatin: Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Hydroxychloroquine: Hydroxychloroquine will be given as a flat dose of 200 mg orally BID (total daily
Period: Overall Study
Arm/Group | Cohort 1: Bevacizumab Eligible Patients | Cohort 2: Bevacizumab Ineligible Patients
Started | 12 | 20
Completed | 0 | 2
Not Completed | 12 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Bevacizumab Eligible Patients | Cohort 2: Bevacizumab Ineligible Patients | Total
Number analyzed (Participants) | 12 | 20 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 3 | 8 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 6 | 12 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 11 | 18 | 29
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 10 | 18 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 20 | 32

OUTCOME MEASURES:

1. Primary Outcome: Antitumor Activity, as Measured by Tumor Response Rate of Hydroxychloroquine, Paclitaxel, Carboplatin, and Bevacizumab (for Eligible Patients) in Patients With Advanced or Recurrent NSCLC Cancer
Description: Assessed using RECIST criteria. Determined using a Simon's two-stage minimax design with a 5% significance level and 80% power.
Time Frame: 6 years
Population: The analysis is comprise of evaluable patients who had measurable disease and received at least one cycle of therapy and had disease evaluated.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Cohort 2: Bevacizumab Ineligible Patients: Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Hydroxychloroquine 200 mg PO BID
  Paclitaxel: Paclitaxel was given at a dose of 200 mg/m2(by IV over 3 hours on Day 1).
  Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Carboplatin: Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Hydroxychloroquine: Hydroxychloroquine will be given as a flat dose of 200 mg orally BID (total daily)
- Cohort 1: Bevacizumab Eligible Patients: Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Bevacizumab 15 mg/kg IV over 90 min for Hydroxychloroquine 200 mg PO BID
  Paclitaxel: Paclitaxel was given at a dose of 200 mg/m2(by IV over 3 hours on Day 1).
  Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Carboplatin: Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Hydroxychloroquine: Hydroxychloroquine 600 mg BID
Arm/Group | Cohort 2: Bevacizumab Ineligible Patients | Cohort 1: Bevacizumab Eligible Patients
Number analyzed (Participants) | 11 | 15
percentage of participants | 55 [23.4 to 83.0] | 27 [7.8 to 55.1]
Statistical Analysis 1: Comparison: Cohort 2: Bevacizumab Ineligible Patients vs Cohort 1: Bevacizumab Eligible Patients; The analysis is comprised of evaluable patients who had measureable disease and received at least one cycle of therapy and had disease evaluated; Test type: Other; p = 0.01, t-test, 2 sided; Mean Difference (Net) = 56, 95% CI 2-sided [8.9 to 72]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Kaplan-Meier estimates of survival were calculated. The median survival times and 95% confidence intervals are presented.
Time Frame: 6 years
Population: Median PFS (in months) were calculated
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cohort 2: Bevacizumab Ineligible Patients: Paclitaxel 200mg/m2 IV over 3 hours Carboplatin AUC= 6 IV over 15-30 min Hydroxychloroquine 200 mg PO BID
  Paclitaxel: Paclitaxel was given at a dose of 200 mg/m2(by IV over 3 hours on Day 1).
  Cycles every 3 weeks for 4-6 Cycles.
  Prior to receiving paclitaxel, all patients will receive the following premedication:
  * Dexamethasone 20 mg po 12 and 6 hours prior to paclitaxel infusion (patients may be treated with dexamethasone 20 mg iv < 1 hour prior to infusion with paclitaxel if the patient did not take the oral dexamethasone)
  * Diphenydramine 50 mg iv (or equivalent) < 1 hour prior to paclitaxel infusion
  * Ranitidine 50 mg iv < 1 hour prior to paclitaxel infusion (alternatively other H2-blockers may be used)
  Carboplatin: Carboplatin will be given at AUC = 6 by IV over 15-30 minutes on Day 1 immediately following paclitaxel. Cycles every 3 weeks for 4-6 Cycles.
  Hydroxychloroquine: Hydroxychloroquine will be given as a flat dose of 200 mg orally BID.
Arm/Group | Cohort 2: Bevacizumab Ineligible Patients | Cohort 1: Bevacizumab Eligible Patients
Number analyzed (Participants) | 11 | 15
months | 4.2 [1.8 to 6.4] | 2.9 [2.0 to 4.6]

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 275 days per patient.
Arm/Group | Cohort 1: Bevacizumab Eligible Patients | Cohort 2: Bevacizumab Ineligible Patients
All-Cause Mortality (participants affected / at risk) | 0/12 | 3/20
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/20
Other Adverse Events (participants affected / at risk) | 0/12 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT01649947/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT01649947/SAP_001.pdf